CLINICAL TRIAL: NCT05906498
Title: Evaluation of the Effect of Acetylcysteine and Vitamin E on Psoriasis Vulgaris Patients During The Active Phase
Brief Title: Using Acetylcysteine and Vitamin E With Psoriasis Vulgaris
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Naira abbas hassan Elkalla, teaching assistant of clinical pharmacy department at BUC, Badr University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Acetylcysteine in Psoriasis
Record Dates: First submitted 2023-06-04; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — Acetylcysteine; Vitamin E

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mix acetylcysteine with vitamin E (Active Comparator): Standard treatment for mild psoriasis, plus N acetyl cysteine (600 mg a day) oral effervescent sachet,30 minutes before breakfast Plus, vitamin E (1000 mg) daily, oral soft gelatin capsule for 8 weeks
  Interventions: Drug: Acetyl cysteine; Drug: Vitamin E
- acetylcysteine (Active Comparator): Standard treatment for mild psoriasis, plus N acetyl cysteine (600 mg a day) oral effervescent sachet, 30 minutes before breakfast, for 8 weeks
  Interventions: Drug: Acetyl cysteine
- standard treatment alone (No Intervention): Standard treatment for mild psoriatic patients (topical steroid and salicylic acid

INTERVENTIONS:
Drug: Acetyl cysteine — N-acetyl cysteine (NAC) is synthetic cysteine amino acid, which in turn elevate the glutathione level in the body, which have important direct antioxidant activity.
  Arms: acetylcysteine; mix acetylcysteine with vitamin E
Drug: Vitamin E — vitamin E possessing an anti-inflammatory action
  Arms: mix acetylcysteine with vitamin E

SUMMARY:
This study aims to assess the effect of adding N-acetyl cysteine (NAC) alone or in combination with Vitamin E to conventional therapy in improving the clinical outcome, oxidative stress, and inflammation in patients with mild psoriasis vulgaris

DETAILED DESCRIPTION:
The study will include 60 Mild psoriatic patients in the active phase (score <, =3) using PASI score. The PASI is a widely used instrument that assesses and grades the severity of psoriatic lesions and the patient's response to treatment. They will assigned randomly into 3 groups. Each group will contain 20 patients. the first group will receive Standard treatment for mild psoriatic patients (topical steroid and salicylic acid), the second group will receive Standard treatment for mild psoriasis, plus N acetyl cysteine (600 mg a day) oral, 30 minutes before breakfast, for 8 weeks. the third group will receive Standard treatment for mild psoriasis, plus N acetyl cysteine (600 mg a day) oral effervescent sachet,30 minutes before breakfast Plus, vitamin E (1000 mg) daily, oral soft gelatin capsule for 8 weeks.

PASI=Psoriasis Area and Severity Index

ELIGIBILITY:
Inclusion Criteria:

1. Adult Patients from 18 to 65 years.
2. Gender: both males and females.
3. Mild psoriatic patients in the active phase (score < =3)
4. Patients diagnosed with mild psoriasis in the active phase (score less than or equal 3) using PASI score.

Exclusion Criteria:

1. Inactive psoriasis vulgaris patients.
2. Alcohol consumption
3. Any other autoimmune diseases.
4. Pregnant or lactating women.
5. Patients with serious illness and any systemic failure (cardiovascular, renal, or respiratory)
6. Patients with major psychiatric or mental illness.
7. Intake of any antioxidants in the previous 3 months
8. Patients of chronic diseases, like hypertension, heart problems
9. Patients with history of bleeding, ulcers, or uncontrollable heartburn.
10. Patients taking anticancer medications that can aggravate psoriasis vulgaris such as mercaptopurine, vinblastine, actinomycin, and Radiation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
level of interleukin-36(IL-36 gamma) (Pg/ml) | 4 months
  measuring level of interleukin-36(IL-36 gamma) at baseline before the intervention and during taking the intervention and 1 month after stopping taking the intervention
level of Malondialdehyde (MDA) (µmol/L) | 4 months
  measuring level of malondialdehyde (MDA) at baseline before the intervention and during taking the intervention and 1 month after stopping taking the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Haud Al-Marsoud Hospital, Cairo, Egypt

REFERENCES:
- [Background] D'Erme AM, Wilsmann-Theis D, Wagenpfeil J, Holzel M, Ferring-Schmitt S, Sternberg S, Wittmann M, Peters B, Bosio A, Bieber T, Wenzel J. IL-36gamma (IL-1F9) is a biomarker for psoriasis skin lesions. J Invest Dermatol. 2015 Apr;135(4):1025-1032. doi: 10.1038/jid.2014.532. Epub 2014 Dec 19. PMID 25525775
- [Background] Yildirim M, Inaloz HS, Baysal V, Delibas N. The role of oxidants and antioxidants in psoriasis. J Eur Acad Dermatol Venereol. 2003 Jan;17(1):34-6. doi: 10.1046/j.1468-3083.2003.00641.x. PMID 12602965
- [Background] Rizvi S, Raza ST, Ahmed F, Ahmad A, Abbas S, Mahdi F. The role of vitamin e in human health and some diseases. Sultan Qaboos Univ Med J. 2014 May;14(2):e157-65. Epub 2014 Apr 7. PMID 24790736